CLINICAL TRIAL: NCT04566991
Title: Deferoxamine In the Treatment of Aneurysmal Subarachnoid Hemorrhage (DISH)
Brief Title: Deferoxamine In the Treatment of Aneurysmal Subarachnoid Hemorrhage (aSAH)
Acronym: DISH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aditya S. Pandey, MD (Other)
Responsible Party: Sponsor-Investigator, Aditya S. Pandey, MD, Associate Professor of Neurosurgery and Associate Professor of Radiology, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00163868
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: Deferoxamine; Placebo
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Deferoxamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: All patients and investigators who will be directly involved in the care of these patients or in data analysis will be blinded to randomization status.This trial uses a Bayesian adaptive randomization protocol, where there are three groups that patients will be randomized into: placebo, DFO 32 mg/kg and DFO 48 mg/kg. The first 50 patients will be randomized evenly into each of these groups. The randomization ratio will be adjusted based on the design report after 50 subjects and then every 10 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Deferoxamine lower dose (Experimental): Deferoxamine 32 Milligram Per Kilogram (mg/kg)
  Interventions: Drug: Deferoxamine
- Deferoxamine higher dose (Experimental): Deferoxamine 48 mg/kg
  Interventions: Drug: Deferoxamine
- Placebo (Placebo Comparator): normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Deferoxamine — There will be 3 doses given to the patients days 1-3. Dose will be given intravenous with a fixed rate of 7.5 milligram per kilogram per hour (mg/kg/hr). The second dose will be given 24 hours after the first dose, and the third dose will be given 48 hours after the initial dose.
  Patients will be randomized to 32 mg/kg or 48 mg/kg of Deferoxamine.
  Other Names: Desferal
  Arms: Deferoxamine higher dose; Deferoxamine lower dose
Drug: Placebo — There will be 3 doses given to the patients days 1-3. Dose will be given intravenous with a fixed rate of 7.5 mg/kg/hr. The second dose will be given 24 hours after the first dose, and the third dose will be given 48 hours after the initial dose.
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
Aneurysmal subarachnoid hemorrhage (aSAH) has a high incidence of mortality and significant morbidity, with mortality exceeding 30% in the first two days.The initial injury is related to increasing intracranial pressure, cerebral edema, and neuronal injuries associated with the release of iron. Iron has been shown to increase the incidence of cerebral edema, ischemia, and formation of hydrocephalus. Deferoxamine mesylate (DFO), a hydrophilic chelator, creates a stable complex with free iron thus preventing the formation of iron related free radicals.

This trial will evaluate the safety and efficacy of clinical deferoxamine for the treatment of aSAH for patients that are admitted to the hospital at the University of Michigan. Eligible participants will be enrolled and randomized to 1 of 2 doses of Deferoxamine or placebo (saline). Information regarding the patients will be collected and followed for up to 6 months post discharge.

ELIGIBILITY:
Inclusion Criteria:

* Aneurysmal SAH confirmed with vascular imaging
* Aneurysm treated with endovascular or microsurgical intervention
* Hunt-Hess ≤ 4
* Modified Fisher Grade I-IV
* Glasgow Coma Scale (GCS) ≥ 7 following External Ventricular Drain (EVD) placement if indicated
* First dose of drug can be administered within 24 hours of symptom onset
* Functional independence prior to SAH, Modified Rankin Scale (mRS) ≤ 1
* Informed consent obtained by patient or legal authorized representative (LAR)

Exclusion Criteria:

* Previous hypersensitivity to or treatment with deferoxamine
* Presence of giant aneurysm (>25 mm in size)
* Known severe iron deficiency anemia, Hemoglobin (Hgb) g/dl ≤ 7 or transfusion dependent
* Irreversibly impaired brainstem function
* Abnormal renal function, Serum Creatinine> 2 mg/dL
* Pre-existing severe disability, mRS ≥ 2
* Coagulopathy, including use of anti-platelet or anticoagulant drugs
* Known severe hearing loss
* Chronic pulmonary disease that limits basic activities of daily living at baseline, or requires the use of home oxygen.
* Acute pulmonary disease with the need for any of the following - in a 72 hour period prior to enrollment: >4L/minute nasal cannula (or equivalent O2 delivery via face mask/ tent), heated-high flow nasal cannula, noninvasive positive pressure ventilation, and in intubated patients FiO2>45% or positive end-expiratory pressure (PEEP) > 8cmH2O. This does not include the use of supplemental oxygen in any form for pre-oxygenation, apneic oxygenation, or peri-procedural support alone.
* Taking iron supplements containing > 325 mg of ferrous iron
* Pregnancy or nursing
* Life expectancy less than 90 days due to co-morbidities
* Concurrent participation in another research protocol for investigation of another experimental therapy, though observational studies are allowed
* Prior history of hepatic dysfunction
* Known cytopenia (platelets < 50,000, Absolute neutrophil count < 500)
* Current use of prochlorperazine
* History of severe psychiatric disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-20 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Utility-weighted modified Rankin Scale (UW-mRS) at 6 months | 6 months (after hospital discharge)
  Overall a Bayesian, longitudinal model will be used, this will be adjusted for baseline expected 6 month mRS using the FRESH score. At baseline, the expected 6 month UW-mRS (based on prognostic variables such as age and Hunt Hess) will be entered as the first value for the patient. Therefore, patients with greater severity at baseline, who achieve excellent outcomes will contribute a larger treatment effect. Similarly, patients with greater severity who have disability, but perform better than expected can still contribute useful information.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MOCA) | At discharge from hospital (approximately 3-4 weeks)
  Montreal cognitive assessment is a rapid sensitive screening tool for assessment of impaired cognitive function. The main domains of MoCA scale include attention, executive functions, memory, language, attention, naming, orientation, and visual-spatial ability. The total score is 30 points. A score of 25 points or less indicated impaired cognitive function. For patients with less than 12 years of education, one point was added to the total score.
Montreal Cognitive Assessment (MOCA) | 6 months (after hospital discharge)
  Montreal cognitive assessment is a rapid sensitive screening tool for assessment of impaired cognitive function. The main domains of MoCA scale include attention, executive functions, memory, language, attention, naming, orientation, and visual-spatial ability. The total score is 30 points. A score of 25 points or less indicated impaired cognitive function. For patients with less than 12 years of education, one point was added to the total score.
Percentage of patients requiring permanent cerebrospinal fluid (CSF) diversion due to hydrocephalus at 6 months | 6 months
Partial pressure of oxygen (PaO2) and fraction of inspired oxygen (FiO2) ratio (worst value for each parameter for each day of infusion, and 48 hours after end of infusion) | up to 48 hours after day 3 infusion
  Worst value for each parameter for each day of infusion, and 48 hours after end of infusion.
To estimate the proportion of non-intubated participants at each dose who experience intubation or initiation of non-invasive positive pressure ventilation during the DFO | infusion days 1-3
Incidence of delayed cerebral ischemia/vasospasm | up to 14 days after aSAH
  This is based on radiographic evidence on computed tomography angiogram and clinical correlation with neurologic exam.

CONTACTS AND LOCATIONS:
Overall Officials: Aditya Pandey, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No